CLINICAL TRIAL: NCT06393725
Title: A Non-Inferiority Trial Comparing Synchronous and Asynchronous Remotely Delivered Lifestyle Interventions
Brief Title: Synchronous vs Asynchronous Remotely Delivered Lifestyle Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H23-0383
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asynchronous (Experimental): This arm involves a 1 year behavioral weight loss program delivered in private Facebook groups led by a professional weight loss counselor. At the end of 1 year, volunteer participants will take over the leadership role of the group for the following year. Volunteers will receive a brief training on how to lead a private Facebook group.
  Interventions: Behavioral: Asynchronous Remote Lifestyle Intervention
- Synchronous (Active Comparator): This arm involves a 1 year behavioral weight loss program delivered via weekly videoconference meetings led by a professional weight loss counselor. At the end of 1 year, volunteer participants will take over the leadership role of the meetings for the following year. Volunteers will receive a brief training on how to lead videoconference meetings.
  Interventions: Behavioral: Synchronous Remote Lifestyle Intervention

INTERVENTIONS:
Behavioral: Asynchronous Remote Lifestyle Intervention — A 1 year lifestyle intervention based on the Diabetes Prevention Program to be delivered asynchronously via a private Facebook group led by a professional weight loss counselor. In the subsequent year, a Peer-Led Maintenance Phase will occur in which a participant volunteer will lead the group after receiving a brief training.
  Arms: Asynchronous
Behavioral: Synchronous Remote Lifestyle Intervention — A 1 year lifestyle intervention based on the Diabetes Prevention Program to be delivered synchronously via weekly videoconference group meetings led by a professional weight loss counselor. In the subsequent year, a Peer-Led Maintenance Phase will occur in which a participant volunteer will lead the group after receiving a brief training.
  Arms: Synchronous

SUMMARY:
The goal of this clinical trial is to learn if a group-based digital weight loss program that is delivered asynchronously (via an online platform) is as effective as one that is delivered synchronously (via weekly videoconference meetings). In the asynchronous condition, participants can engage with their group any time 24/7. In the synchronous condition, participants can engage with their group once a week at a videoconference meeting. The main questions it aims to answer are:

Will participants in each condition lose about the same amount of weight? Will the participants in the asynchronous condition participate more than those in the synchronous condition? Will the participants in the asynchronous condition feel more connected to each other than those in the synchronous condition? Will the asynchronous condition cost less to deliver per pound lost than the synchronous condition?

Participants will:

Receive a digital weight loss program that lasts 1 year and then volunteer participants will be selected to lead the group for 1 year following the program, a phase called the "peer-led weight loss maintenance phase." Complete study assessments at baseline, 6, 12, 18, and 24 months.

DETAILED DESCRIPTION:
Lifestyle interventions have had established efficacy for decades but they are costly and have poor scalability. Remotely-delivered lifestyle interventions have increased the potential for scale and systematic reviews have found that they are effective, especially those that include human coaching. Some remote lifestyle interventions are synchronous, such that they are delivered via videoconferencing or phone. Other remote lifestyle interventions are asynchronous, such that they are delivered via online platforms that allow for clinicians and patients to engage via text exchanges or via online groups where patients engage with a clinician and each other by posting messages and contributing to discussion threads. The advantage of asynchronous approaches are 24/7 accessibility which makes them conducive to "just in time" support, allowing patients to engage anytime they want to, as opposed to in scheduled blocks of time each week. Asynchronous, remote interventions may also be more scalable than synchronous remote interventions. A trial of two asynchronous, remote lifestyle interventions-one with a group of 94 participants and one with a group of 40 participants revealed similar weight loss and acceptability between conditions. The larger group was also more sustainable, such that participants continued to engage in the group for longer when the groups were turned over to participants to lead themselves for a year after the intervention ended-a period referred to as the peer-led maintenance phase. The next step in this research is to examine how an asynchronous, remote intervention compares to a synchronous, remote intervention, not only in short term weight loss, but also in sustainability, scalability, and weight loss maintenance. Now that the feasibility of conducing large asynchronous, remote groups has been established, the proposed trial will randomize participants to large groups (n=82) in both conditions, which will allow the comparison of synchronous to asynchronous remote interventions that are scaled up to a level established as acceptable for asynchronous remote interventions. The purpose of the proposed trial is to determine whether an asynchronous, remote lifestyle intervention is non-inferior to a synchronous, remote lifestyle intervention in weight loss at 6 and 12 months, but more scalable and sustainable, and thus producing greater weight loss maintenance at 18 and 24 months. Establishing evidence for asynchronous interventions is more important than ever given that telehealth reimbursement for behavioral health has recently expanded but is still limited to synchronous forms of remote care. Asynchronous interventions may be more convenient for some people and possibly more scalable but for this treatment model to reach its potential, evidence for efficacy is needed to inform reimbursement policy. The hypothesis is that an asynchronous, remote lifestyle intervention will produce similar initial weight loss as a synchronous, remote version but will be less expensive, more sustainable, and generate greater collective efficacy, which will drive greater weight loss maintenance at 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-45
* has Bluetooth or wifi connectivity at home (for scale)
* goes on Facebook at least 5 days per week over the past 2 weeks
* has posted/replied at least once a week in the past 2 weeks (per self-report)
* has a smart phone

Exclusion Criteria:

* Pregnant or lactating or plans to during study period
* bipolar disorder, substance abuse, psychosis, bulimia, binge eating disorder, or severe depression
* had bariatric surgery or plans to during the study
* currently taking meds affecting weight
* lost ≥5% of weight in past 6 months
* participating in another weight loss program or plans to during the study
* chronic pain or medical condition that interferes with the ability to exercise
* type 1 diabetes
* unable to walk ¼ mile unaided without stopping
* nicotine user

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent of baseline weight loss at 6 months | 6 months
  Percent weight loss
Percent of baseline weight loss at 12 months | 12 months
  Percent weight loss

SECONDARY OUTCOMES:
Word count of participant engagement in 1 year | 1 year
  word count
Word count of participant engagement in 2 years | 2 years
  word count
Collective Efficacy | 1 year
  Online Collective Efficacy Scale score out of a range of 0-210 where higher scores indicate greater collective efficacy
Collective Efficacy | 2 years
  Online Collective Efficacy Scale score out of a range of 0-210 where higher scores indicate greater collective efficacy
Cost in dollars per pound lost | 1 year
  Intervention cost will be computed for each participant and then divided by pounds lost
Cost in dollars per pound lost | 2 years
  Intervention cost will be computed for each participant and then divided by pounds lost
Percent of baseline weight lost at 18 months | 18 months
  Percent weight loss
Percent of baseline weight lost at 24 months | 24 months
  Percent weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Pagoto, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
The data and associated documentation will be made available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Datasets will be stored with encryption and will be shared only after verification of human subjects institutional review board approval is obtained. By requesting human studies approval, we will be able to track recipients of the data, the type of data analyses proposed, and subsequent research findings. All storage and sharing of data will be in accordance with the policy and approval of University of Connecticut institutional review board.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available 1 year following the end of the trial. It will be available for 5 years.
Access Criteria: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Pagoto S, Xu R, Bannor R, Idiong C, Goetz J, Fernandes D. Comparing Synchronous and Asynchronous Remotely Delivered Lifestyle Interventions: Protocol for a Randomized Noninferiority Trial. JMIR Res Protoc. 2024 Dec 19;13:e65323. doi: 10.2196/65323. PMID 39700497

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT06393725/Prot_SAP_000.pdf